CLINICAL TRIAL: NCT06520501
Title: Comparison of the Effectiveness of Sambiloto Herbs (Andrographis Paniculata) and Brisk Walking Exercise on Blood Glucose of Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Palangka Raya (Other)
Responsible Party: Principal Investigator, Agnes Veronica Agustin, Ketua Komite Etik, Universitas Palangka Raya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2504031946
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: MeSH
Keywords: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Brisk Walking (Experimental): Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.
  Interventions: Behavioral: Brisk Walking
- Herbal Medicine Sambiloto (Experimental): Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Interventions: Dietary Supplement: Herbal Medicine Sambiloto
- Combination (Experimental): Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.
  Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Interventions: Combination Product: Brisk Walking and Herbal Medicine Sambiloto
- Control Obese (No Intervention): Obese with no intervention
- Control Normal (No Intervention): Normal with no intervention

INTERVENTIONS:
Dietary Supplement: Herbal Medicine Sambiloto — Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days.
  Arms: Herbal Medicine Sambiloto
Behavioral: Brisk Walking — Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute.
  Arms: Brisk Walking
Combination Product: Brisk Walking and Herbal Medicine Sambiloto — Moderate activity that uses brisk walking techniques for 30 minutes at an average speed of up to 5 km/h or 100 steps per minute. Jamu Sambiloto is herbal medicine obtained through products that already have a distribution permit and have a distribution permit registration number, with a consumption dose of 1 capul / day or 350 grams for 7 consecutive days
  Arms: Combination

SUMMARY:
Problem Formulation

1. Does herbal medicine sambiloto affect the blood glucose levels of obese sufferers?
2. Does brisk walking affect blood glucose levels in obese sufferers?
3. Does the combination of bitter herbal medicine and brisk walking have an effect on blood glucose levels in obese sufferers?
4. Is there a difference in the effectiveness between herbal bitter and brisk walking and the combination on blood glucose levels in obese sufferers?

Research Objectives

General Objectives :

The general aim of this research is to determine the difference in effectiveness between the herbal medicine Sambiloto and brisk walking as well as the combination on the blood glucose levels of obese sufferers.

Specific Objective :

1. Knowing the effect of herbal medicine Sambiloto on blood glucose in obese sufferers.
2. Knowing the effect of brisk walking on blood glucose in obese sufferers.
3. To determine the effect of the combination of herbal medicine Sambiloto and brisk walking on blood glucose levels in obese sufferers.

DETAILED DESCRIPTION:
This type of research uses the Quasi Experimental method type Non-equivalent control group design, with a research design in the form of two group pre test and post test design, in this study there are two groups that will be measured pretest before intervention and post test after intervention and 1 control group without being given intervention. The intervention group is divided into two groups, namely the group given the herbal medicine sambiloto, and the group given the Brisk Walking Exercise treatment. Quasi-experimental research design with research design in the form of two group pre test and post test design.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to be a respondent with informed consent
2. Obesity sufferers in the Jekan Raya District area
3. Have a BMI ≥ 25 kg/m2 (Obesity I)
4. Adult age (19-39 years)

Exclusion Criteria:

1. Not being present or out of town during the research
2. Unable to continue research due to serious illness or death
3. Withdraw while participating in the research
4. Have a history of drug allergies
5. Experiencing decreased consciousness
6. Experiencing an extremity injury
7. Have a history of cardiovascular disease, kidney disease or stomach ulcers
8. Have a history of bloody stools
9. Are pregnant or breastfeeding

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-04 (Estimated); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Differences | 7 consecutive day
  Difference in blood glucose before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Veronica Agustin, Principal Investigator — Universitas Palangka Raya

IPD SHARING:
Plan to Share IPD: Undecided